CLINICAL TRIAL: NCT03400592
Title: Multi-center Phase II Trial of Nimotuzumab Plus Irinotecan in Patients With High EGFR Expression After Failure of First-line Treatment in Recurrent or Metastatic Gastric Adenocarcinoma（NIEGA）
Brief Title: Study of Nimotuzumab and Irinotecan as Second Line With Recurrent or Metastatic Gastric Adenocarcinoma
Acronym: NIEGA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Shen Lin, Head of Department of GI oncology, Beijing Cancer Hospital, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIEGA
Record Dates: First submitted 2015-10-10; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Stomach Neoplasms
Keywords: gastric adenocarcinoma; EGFR; Irinotecan; Nimotuzumab; biomarker
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan; nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- irinotecan and nimotuzumab (Experimental): Administration of irinotecan 180 mg/m2 IV once every 2 weeks and nimotuzumab 400 mg IV once weekly
  Interventions: Drug: Irinotecan; Drug: nimotuzumab

INTERVENTIONS:
Drug: Irinotecan — 180 mg/m2 IV once every 2 weeks until radiographically documented tumour progression, unacceptable toxicity, or withdrawal of consent by the patient
Drug: nimotuzumab — 400mg IV once weekly until radiographically documented tumour progression, unacceptable toxicity, or withdrawal of consent by the patient

SUMMARY:
The trial aims to evaluate the efficacy and safety of adding nimotuzumab to irinotecan after failure of first-line treatment in recurrent or metastatic gastric adenocarcinoma with overexpression of EGFR, and search for the effective biomarkers for nimotuzumab efficacy in gastric cancer.

DETAILED DESCRIPTION:
The sample size was calculated using Simon's 2-stage design. The first stage require at least 4 or more out of 19 patients to have a confirmed partial or complete response (assuming P1 = 0.30, P0 = 0.10, with alpha = 0.05 and beta = 0.2) before proceeding to the second stage, in which additional 36 patients were needed. If a total of 15 or more patients achieve a confirmed objective response, then the primary end-point would have been met. The predicted response rate in this study is at least 30%. Blood and tissue samples are required to collect at baseline, response and disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Advanced unresectable or recurrent gastric or gastroesophageal junction adenocarcinoma patients which meet the following criteria:
* Willing to sign ICF
* Above 18 years
* KPS score≥70
* Expected survival time more than 90 days
* Subjects with EGFR overexpression (2+ or 3+ in IHC)
* With target lesions in spiral CT or MRI examination within 30 days
* Subjects who experienced disease progression during first line or within 6 months after the last dose of first line therapy. The first line regimen must have contained a 5-fluorouracil based agent ,platinum agent and Paclitaxel agent.
* Lab test of baseline meet following criteria
* Hemoglobin higher than 9.0g/dL
* Neutrophil higher than 1,500/mm3
* PLT higher than 10.0 104/mm3
* Bilirubin lower than 1.5 times of upper limit of normal range
* AST,ALT,ALP lower than 2.5 times of upper limit of normal range
* Creatinine lower than upper limit of normal range
* When patient has liver metastasis or bone metastasis, the value of AST,ALT,ALP could be within 5 times of upper limit of normal range

Exclusion Criteria:

* Patients who have received irinotecan
* Patients who are allergic to irinotecan or nimotuzumab.
* Other active malignancy within the last 5 years
* Female patients who are in pregnancy or lactation and patients who are not willing to take contraception measures
* Investigator judge not eligible to this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  CT/MRI will be performed every 2 cycles of treatment by RECIST 1.1.Overall Response Rate is defined as the proportion of subjects with CR or PR in the best overall response

SECONDARY OUTCOMES:
Overall survival | 3 years after first enrollment
  Overall survival is defined as the time from the date of enrollment to the date of the death from any cause.
Progression free survival | 3 years after first enrollment
  Progression Free Survival is defined as the time from the date of enrollment to the date of progression or death from any cause
Disease control rate | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Disease Control Rate is defined as the proportion of subjects with CR, PR or SD in the best overall response
Safety | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Potential predictive biomarkers of nimotuzumab | 3 years after first enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Peking cancer hospital, Beijing, Beijing Municipality, China